CLINICAL TRIAL: NCT04084795
Title: Augmentation of EMDR With Transcranial Direct Current Stimulation (tDCS) in the Treatment of Fibromyalgia: a Double-blind Randomized Controlled Trial
Brief Title: Augmentation of EMDR With tDCS in the Treatment of Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Universitat Oberta de Catalunya (Other)
Responsible Party: Principal Investigator, Alicia Valiente, Principal investigator, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019/8772/I
Record Dates: First submitted 2019-08-02; First posted 2019-09-10 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Fibromyalgia; Psychological Trauma; Depressive Symptoms; Anxiety
Keywords: Fibromyalgia; Psychological trauma; Posttraumatic stress disorder; Major depressive disorder; Anxiety disorder; Eye Movement Desensitization and Reprocessing; transcranial Direct Current Stimulation
MeSH Terms: conditions — Fibromyalgia; Psychological Trauma; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Depressive Disorder, Major | interventions — Eye Movement Desensitization Reprocessing; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant and the care provider will be blind to the tDCS condition as sham-tDCS will be used, whereas the Outcomes assessor will be blind to both conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- EMDR plus tDCS (Active Comparator): tDCS stimulation will consist of 2mA tDCS for 20 minutes applied immediately before EMDR sessions.
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing therapy; Other: transcranial Direct Current Stimulation
- EMDR plus sham-tDCS (Placebo Comparator): Sham stimulation will consist of inactive tDCS for 20 minutes applied immediately before EMDR sessions
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing therapy
- Treatment as Usual (No Intervention): Patients in this condition will not receive EMDR nor tDCS sessions, and will continue to attend their regular visits with rheumatology and psychiatry.

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing therapy — EMDR is a psychotherapeutic approach using a standardized 8-phase protocol to alleviate the distress associated with traumatic memories, facilitating the access to and processing of traumatic memories. Patients will receive 20 individual EMDR sessions of 60 minutes each using the standard protocol, as well as a specific pain protocol and the fibromyalgia protocol. EMDR is an integrative psychotherapy that uses standardized protocols and elements of cognitive-behavioral, interpersonal, and body-centered therapies, as well as dual stimulation (e.g., side-to-side eye movements).
  The current standard protocol includes eight phases:
  Patient history. Patient preparation. Patient assessment. Memory desensitization. Installing the positive cognition. Body scan. Closure. Reevaluation.
  Other Names: EMDR
  Arms: EMDR plus sham-tDCS; EMDR plus tDCS
Other: transcranial Direct Current Stimulation — tDCS represents a promising intervention option, given its capacity to modulate cerebral excitability in a simple, safe manner. F3 anodal; Fp1, F7, Fc5, AF3, Fc1, Fz, return montage will be used with the anode over the left DLPFC. Half of the patients will receive active stimulation and the other half sham stimulation. Active stimulation will consist of 2mA tDCS for 20 minutes applied immediately before EMDR sessions. The same protocol and montage will be used for sham stimulation.
  Other Names: tDCS
  Arms: EMDR plus tDCS

SUMMARY:
Fibromyalgia (FM) is a generalized, widespread chronic pain disorder and has an estimated prevalence of 2%-4% in the general population. Current pharmacological and psychological interventions frequently produce limited benefits in FM patients. Due to FM's strong association with psychological trauma causing neurobiological alterations in stress response, a trauma-focused psychotherapy is an innovative alternative treatment option. Eye Movement Desensitization and Reprocessing (EMDR) has been recognized by the World Health Organization as a first-line therapeutic tool for post-traumatic stress disorder and first evidence suggests that it is also beneficial for patients with FM. Given the complex etiology of FM, a combination of psychotherapy with other treatment options can maximize a potential therapeutic success. A possible candidate herby is transcranial Direct Current Stimulation (tDCS), a non-invasive stimulation technique, which can modify neural activities related to pain and which has shown short-term positive effects on chronic pain and quality of life in FM patients. The patient sample will consist of 96 female patients meeting 2016 American College of Rheumatology criteria for FM based on a clinical interview. They will be randomized to 20 sessions of EMDR plus tDCS or EMDR plus sham-tDCS, or Treatment as Usual (TAU). Therapists, raters, and patients will be kept blind to tDCS treatment conditions. Evaluations will be at baseline, post treatment at 6 months, and follow-up at 12 months. Hypotheses are that EMDR improves pain intensity and clinical symptoms at short and long-term, and that tDCS enhances this effect, which will be superior to tDCS-sham.

DETAILED DESCRIPTION:
Fibromyalgia (FM) affects 2-4% of the general population with typical symptoms such as generalized and widespread pain, sleep disturbances, problems in memory and attention, anxiety and depression. Pharmacological treatment and psychotherapeutic interventions have produced limited effects so far. Interestingly, lifetime psychosocial adversities are substantially elevated in FM but no interventions are currently offered. Given the complex etiology of FM, combining a psychotherapy with other treatment options can maximize the potential benefit of this intervention. The investigators will test in Barcelona, whether a trauma-oriented therapy, Eye Movement Desensitization Reprocessing (EMDR), in combination with a non-invasive brain stimulation technique, transcranial Direct Current Stimulation (tDCS), can improve typical FM symptoms.

Outcomes

Primary outcomes:

1. To test whether EMDR plus tDCS or EMDR plus sham-tDCS in comparison to TAU group, improve pain intensity, depressive and anxious symptoms and trauma associated symptoms after therapy and follow-up.
2. To test whether an improvement in pain intensity, depressive and anxious symptoms and trauma associated symptoms can be augmented by simultaneous tDCS comparing EMDR plus tDCS with EMDR plus sham-tDCS after the intervention and whether this is maintained at the follow-up visit.

   Secondary outcomes:
3. To test whether the EMDR plus tDCS or EMDR plus sham-tDCS in comparison to TAU group, improves more in subjective wellbeing after the treatment, and whether this is maintained at the follow-up visit.

Indicators to monitor clinical changes will be performed via various standard self- and hetero-applied scales by blind-to-treatment raters and information provided by patients and the medical chart IT system of our catchment area at baseline (visit 1), post treatment at 6 months (visit 2), and follow-up evaluation at 12 months (visit 3).

This multicenter collaborative project will involve the participation of the Psychiatric Department of the Parc de Salut Mar responsible for coordinating the study, the Rheumatology Department of the Parc de Salut Mar responsible for patient recruitment, and the Cognitive Neuro-Lab of the Universitat Oberta de Catalunya for guidance and council on tDCS use.

Design

Within a double-blind randomized controlled design, patients will be randomized to one of the following three treatment arms:

EMDR with tDCS (20 sessions) vs EMDR with sham-tDCS (20 sessions) vs TAU. Psychotherapists, raters, and patients will be kept blind for tDCS treatment conditions until the end of the trial.

Participants

The patient sample will consist of 96 females fulfilling the 2016 American College of Rheumatology criteria for FM based on clinical interview (Wolfe et al, 2010).

Interventions

* EMDR therapy
* transcranial Direct Current Stimulation (tDCS)
* Treatment as Usual

Randomizations

Participants were randomly assigned to one of the three study groups using REDCap's stratified randomization module to ensure balanced allocation in terms of Revised Fibromyalgia Impact Questionnaire (FIQ-R) score and education level. When a new participant is enrolled, REDCap identifies their stratum based on the data for these two variables, then it assigns them to a study arm using block randomization within that stratum, favoring the arm with the fewest current assignments to maintain balance. The allocation sequence is concealed from outcome raters until participants have finished the trial. This randomization module enforces balance by prioritizing equal group sizes within strata, even with uneven stratum sizes, it provides real-time adaptations by adjusting assignments dynamically as participants enroll and it logs all randomization events for reproducibility purposes.

Computation of sample size

The main tests of the study will consist of assessing whether patients assigned to EMDR show different levels in the pain intensity variable using a standard formula for two-tailed t-tests. The total sample size required to detect large to very large effect size differences (Cohen's d ≥ 1) between three groups with a significance level of 0.05 and statistical power of 80% is 28. Assuming 15% dropouts, we will aim to randomize 96 patients, meaning 32 per group.

Statistical Analysis

The distribution of socio-demographic and clinical characteristics between groups at baseline will be summarized using descriptive statistics. The change in clinical and functional variables from the baseline evaluation to post intervention will be analyzed using linear model t-tests, including as regressors of no interest the potential confounders (age, pain score, anxiety and depression severity, and number of years in education). The statistical software used for the analysis will be the latest available version of R. The investigators will conduct an intention to treat (ITT) analysis, and will use the "Last Observation Carried Forward" (LOCF) method for losses at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old
* Mean pain score of at least 4 on the visual analog scale (VAS) in the two weeks preceding the clinical trial
* Presence of one or more traumatic events causing current trauma-related symptoms
* Current clinical symptoms of depression and/or anxiety
* 2 weeks of stable medication

Exclusion Criteria:

* Comorbid autoimmune or chronic inflammatory disease
* Neurological or serious medical diseases
* Bipolar disorder, schizoaffective disorder and schizophrenia
* Suicidal ideation
* Previous EMDR therapy in the past two years
* Substance abuse/dependency within 1 month prior to participation (except for nicotine abuse/dependency),
* Pending FM-related litigation or disability
* Metallic implants in the head
* Positive test for pregnancy
* Skin sensitivity diseases (psoriasis, eczema, dermatitis, etc.)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The relevance of the current proposal is underscored by a review (Borchers & Gershwin, 2015) on FM, where the authors highlight that it is a frequent disorder with mainly women of low educational level and socio-economic status affected. Moreover, in Spain, the distribution by sex prevalence has been found to be 4.49% in women; significantly higher than the 0.29% in men (Font Gayà et al., 2020).
Enrollment: 96 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in severity and in pain intensity as measured by the Visual Analogue Scale (VAS) | Change from baseline to visits at 6 and 12 months
  The VAS pain consists of a straight horizontal line anchored between 2 verbal descriptors: "No pain" on the left side and "Unbearable pain" on the right. Scores are interpreted as follows: no pain (0-2), mild pain (2-4), moderate pain (4-6), severe pain (6-8), and maximum pain (8-10). This measure assesses the intensity of the perceived pain over the last 2 weeks.
Change in physical impairment due to FM assessed by The Revised Fibromyalgia Impact Questionnaire (FIQ-R) | Change from baseline to visits at 6 and 12 months
  9-item self-administered scale for measuring physical impairment due to FM over the last week. Scores range from 0-100 and higher scores indicate greater impact in functioning.
Change in catastrophic thinking related to pain experiences assessed by the Pain Catastrophizing Scale (PCS) | Change from baseline to visits at 6 and 12 months
  13 item self-report questionnaire designed to assess the extent to which individuals magnify, ruminate, and feel helpless about their pain. Scores range from 0-52 with higher scores indicating greater catastrophizing.
Change in the impact of fatigue as assessed by the Brief Fatigue Inventory (BFI) | Change from baseline to visits at 6 and 12 months
  9 item self-report questionnaire used to assess the severity and impact of fatigue on individuals in the past 24h, as well as its interference with various aspects of daily life, such as mood, walking ability, work, relationships, and enjoyment of life. Scores range from 0-10 with 0: "no fatigue"; 1-3: "low"; 4-6: "moderate" y 7-10: "severe"
PTSD diagnosis assessed by the Global Evaluation of Posttraumatic Stress (EGEP-5) | Change from baseline to 6 and 12 months
  55-item clinician-applied scale to determine current PTSD diagnosis, based on DSM-V criteria. The scale can determine a diagnosis of PTSD, specifying the presence of dissociative symptoms (depersonalization and derealization) and delayed expression.
Complex PTSD diagnosis assessed by The International Trauma Questionnaire (ITQ) | Measure at baseline
  This 12 item questionnaire is a tool used to evaluate and diagnose complex post-traumatic stress disorder (C-PTSD) and other trauma-related disorders, in terms of ICD-11 classification for mental disorders. It assess the presence and severity of PTSD symptoms, as well as disturbances in self-organization associated with C-PTSD.
Change in PTSD symptoms as measured by the Posttraumatic Stress Disorder Checklist (PCL-5) | Change from baseline to visits at 6 and 12 months
  This scale assesses DSM-5 PTSD symptoms using a 20-item questionnaire. Scores range from 0 to 80, with higher scores indicating greater severity. A cut-off score of 33 is used for diagnosis.
Change in subjective perceived distress assessed by Subjective unit of distress (SUD) | Change from baseline to visits at 6 and 12 months
  this scale, ranging from 0 (no distress) to 10 (maximum distress), evaluates the level of subjective perturbation a person experiences when they bring to mind the traumatic event chosen in the EGEP-5 scale.
Quantifying childhood trauma assessed by The Childhood Trauma Questionnaire (CTQ) | Measure at baseline.
  Self-applied scale which includes a 28-item test that measure 5 types of childhood maltreatment: emotional, physical and sexual abuse, and emotional or physical neglect. A 5-point Likert scale (from 1 to 5) is used for the responses which range from "never true" to "very often true". The final scores provide a severity score for each subscale from "none to minimal," "low to moderate," "moderate to severe," and "severe to extreme".
Assessing lifetime trauma with the Timeline of traumatic experiences | Measure at baseline
  The Timeline of traumatic experiences tool was developed specifically for this study and consists of a table that qualitatively compiles different traumatic events that the person may have suffered both in childhood and in adulthood. The table is segmented into 5-year intervals ranging from 0-5 years old to 65-70 years old. Within each segment, participants are asked: "Do you recall experiencing any traumatic or stressful events during this age interval?"
Change in depersonalization symptoms assessed by The Cambridge Depersonalization Scale (CDS) | Change from baseline to 6 and 12 months.
  A self-report questionnaire designed to assess the severity of depersonalization symptoms. It consists of 29 items that evaluate various aspects of depersonalization, including feelings of detachment from oneself, altered perceptions of time and space, and experiences of unreality. Each item on the CDS is rated on two Likert scales: one for frequency and one for duration. The total score ranges from 0 to 290. A higher total score indicates greater severity of depersonalization symptoms with a cut-off point of 70 to indicate depersonalization symptoms.
Change in somatoform dissociation symptoms assessed by Somatoform Dissociation Questionnaire 20 (SDQ-20) | Change from baseline to visits at 6 and 12 months
  The SDQ-20 is a 20-item self-report questionnaire measuring somatoform dissociation. Items refer to somatic symptoms and then ask if there is a known cause for them. The items are answered on a 5-point Likert scale and the symptoms with no known cause are summed to achieve the total scorwhich can range from 20 to 100. A higher score indicates a greater degree of somatoform dissociation.
Change in anxious and depressive symptoms assessed by with the Hospital Anxiety and Depression Scale | Change from baseline to visits at 6 and 12 months
  Severity and changes in anxious and depressive symptoms will be evaluated with the Hospital Anxiety and Depression Scale. Items are rated on a 4-point Likert scale from 0 and 3, yielding a total score ranging from 0 to 21 and a cut-off score of 8 indicating probable clinical symptoms.

SECONDARY OUTCOMES:
Change in subjective wellbeing measured with the Satisfaction With Life Scale. | Change from baseline to visits at 6 and 12 months
  The improvement of subjective wellbeing will be evaluated using the Satisfaction With Life Scale. This scale is completed by 5 items rated from 1 (totally agree) to 5 (totally disagree), with a maximum score of 25.Higher scores mean greater satisfaction.
Change in insomnia symptoms assessed with the Athens Insomnia Scale. | Change from baseline to visits at 6 and 12 months
  The improvement of insomnia symptoms will be evaluated using the Athens Insomnia Scale. This scale is completed by 8 items rated from 0 to 3, with a maximum score of 24. Higher scores mean greater impact of insomnia.
Change in Self-care assessed with The González self-care scale. | Change from baseline to 6 and 12 months.
  This Scale consists of 31 items ona 1 to 7 point Likert scale, grouped into six different components, addressing various aspects of self-care: (1) Self-Destruction: Refers to behaviors that harm us in some way; (2) Lack of Tolerance for Positive Affect: Refers to difficulty in receiving affectionate comments or behaviors from others; (3) Problems in Allowing Help: Refers to difficulty in allowing other people to help us; (4) Resentment for Non-Reciprocity: Refers to the anger felt because our needs or emotions have not been attended to or reciprocated; (5) Lack of Positive Activities: Refers to the absence of activities that make us feel good or are healthy for us; (6) Neglecting One's Own Needs: Refers to the difficulty in identifying and satisfying our own needs. A total score above three on each factor is indicative of dysfunctionality.
Change in emotion regulation assessed with The Emotion-Regulation Skills Questionnaire (ERSQ). | Change from baseline to 6 and 12 months.
  It consists of 27 items that evaluate various emotion-regulation strategies, including cognitive reappraisal, acceptance, problem-solving, and suppression. It is scored on a Likert Scale from 0 to 4, with a total score being the mean. Higher scores indicate greater emotional regulation. The ERSQ provides insight into an individual's skill level in managing their emotions, which can be useful in clinical settings for developing targeted interventions or in research settings for studying emotion regulation across different populations.
Change in self-esteem assessed with The Rosenberg Self-Esteem Scale (RSE). | Change from baseline to 6 and 12 months.
  The RSE consists of ten items that assess an individual's overall feelings of self-worth and self-acceptance. The scale covers both positive and negative aspects of self-esteem, it uses a 4 point Likert scale with higher scores indicating greater levels of self-esteem; from 30 to 40 points: High self-esteem, 26 to 29: average self-esteem, < 25: low self-esteem. The RSE is frequently utilized in research and clinical settings to evaluate self-esteem levels across various populations and to assess the impact of interventions aimed at improving self-esteem.
Change in cognitive function assessed with The Screen for Cognitive Impairment in Psychiatry (SCIP). | Change from baseline to 6 and 12 months.
  The SCIP is a screening tool used to assess cognitive function in psychiatric patients. It consists of a series of brief cognitive tests designed to evaluate various cognitive domains, including memory, attention, executive function, and language. The SCIP is used by mental health professionals to quickly identify cognitive deficits in patients with psychiatric disorders, which can help inform treatment planning and intervention strategies. The total score for the SCIP can range from 0 to 100, with higher scores indicating better cognitive performance.

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt L. Amann, M.D., Principal Investigator — Parc de Salut Mar
Locations (1):
- Centre Forum (Parc de Salut Mar), Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Font Gaya T, Bordoy Ferrer C, Juan Mas A, Seoane-Mato D, Alvarez Reyes F, Delgado Sanchez M, Martinez Dubois C, Sanchez-Fernandez SA, Marena Rojas Vargas L, Garcia Morales PV, Olive A, Rubio Munoz P, Larrosa M, Navarro Ricos N, Sanchez-Piedra C, Diaz-Gonzalez F, Bustabad-Reyes S; Working Group Proyecto EPISER2016. Prevalence of fibromyalgia and associated factors in Spain. Clin Exp Rheumatol. 2020 Jan-Feb;38 Suppl 123(1):47-52. Epub 2020 Jan 8. PMID 31928589
- [Background] Benor D, Rossiter-Thornton J, Toussaint L. A Randomized, Controlled Trial of Wholistic Hybrid Derived From Eye Movement Desensitization and Reprocessing and Emotional Freedom Technique (WHEE) for Self-Treatment of Pain, Depression, and Anxiety in Chronic Pain Patients. J Evid Based Complementary Altern Med. 2017 Apr;22(2):268-277. doi: 10.1177/2156587216659400. Epub 2016 Jul 20. PMID 27432773
- [Background] Bernardy K, Klose P, Busch AJ, Choy EH, Hauser W. Cognitive behavioural therapies for fibromyalgia. Cochrane Database Syst Rev. 2013 Sep 10;2013(9):CD009796. doi: 10.1002/14651858.CD009796.pub2. PMID 24018611
- [Background] Borchers AT, Gershwin ME. Fibromyalgia: A Critical and Comprehensive Review. Clin Rev Allergy Immunol. 2015 Oct;49(2):100-51. doi: 10.1007/s12016-015-8509-4. PMID 26445775
- [Background] Burke NN, Finn DP, McGuire BE, Roche M. Psychological stress in early life as a predisposing factor for the development of chronic pain: Clinical and preclinical evidence and neurobiological mechanisms. J Neurosci Res. 2017 Jun;95(6):1257-1270. doi: 10.1002/jnr.23802. Epub 2016 Jul 12. PMID 27402412
- [Background] Cohen H, Neumann L, Haiman Y, Matar MA, Press J, Buskila D. Prevalence of post-traumatic stress disorder in fibromyalgia patients: overlapping syndromes or post-traumatic fibromyalgia syndrome? Semin Arthritis Rheum. 2002 Aug;32(1):38-50. doi: 10.1053/sarh.2002.33719. PMID 12219319
- [Background] Collado A, Gomez E, Coscolla R, Sunyol R, Sole E, Rivera J, Altarriba E, Carbonell J, Castells X. Work, family and social environment in patients with Fibromyalgia in Spain: an epidemiological study: EPIFFAC study. BMC Health Serv Res. 2014 Nov 11;14:513. doi: 10.1186/s12913-014-0513-5. PMID 25385047
- [Background] Crettaz B, Marziniak M, Willeke P, Young P, Hellhammer D, Stumpf A, Burgmer M. Stress-induced allodynia--evidence of increased pain sensitivity in healthy humans and patients with chronic pain after experimentally induced psychosocial stress. PLoS One. 2013 Aug 7;8(8):e69460. doi: 10.1371/journal.pone.0069460. eCollection 2013. PMID 23950894
- [Background] Hampstead BM, Briceno EM, Mascaro N, Mourdoukoutas A, Bikson M. Current Status of Transcranial Direct Current Stimulation in Posttraumatic Stress and Other Anxiety Disorders. Curr Behav Neurosci Rep. 2016 Jun;3(2):95-101. doi: 10.1007/s40473-016-0070-9. Epub 2016 Mar 28. PMID 29479515
- [Background] Lumley MA, Schubiner H, Lockhart NA, Kidwell KM, Harte SE, Clauw DJ, Williams DA. Emotional awareness and expression therapy, cognitive behavioral therapy, and education for fibromyalgia: a cluster-randomized controlled trial. Pain. 2017 Dec;158(12):2354-2363. doi: 10.1097/j.pain.0000000000001036. PMID 28796118
- [Background] O'Connell NE, Marston L, Spencer S, DeSouza LH, Wand BM. Non-invasive brain stimulation techniques for chronic pain. Cochrane Database Syst Rev. 2018 Mar 16;3(3):CD008208. doi: 10.1002/14651858.CD008208.pub4. PMID 29547226
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] Yavne Y, Amital D, Watad A, Tiosano S, Amital H. A systematic review of precipitating physical and psychological traumatic events in the development of fibromyalgia. Semin Arthritis Rheum. 2018 Aug;48(1):121-133. doi: 10.1016/j.semarthrit.2017.12.011. Epub 2018 Jan 10. PMID 29428291
- [Derived] Gardoki-Souto I, Martin de la Torre O, Hogg B, Redolar-Ripoll D, Martinez Sadurni L, Fontana-McNally M, Blanch JM, Lupo W, Perez V, Radua J, Amann BL, Valiente-Gomez A, Moreno-Alcazar A. The study protocol of a double-blind randomized controlled trial of EMDR and multifocal transcranial current stimulation (MtCS) as augmentation strategy in patients with fibromyalgia. Trials. 2024 Dec 31;25(1):856. doi: 10.1186/s13063-024-08708-3. PMID 39741323
- [Derived] Gardoki-Souto I, Martin de la Torre O, Hogg B, Redolar-Ripoll D, Valiente-Gomez A, Martinez Sadurni L, Blanch JM, Lupo W, Perez V, Radua J, Amann BL, Moreno-Alcazar A. Augmentation of EMDR with multifocal transcranial current stimulation (MtCS) in the treatment of fibromyalgia: study protocol of a double-blind randomized controlled exploratory and pragmatic trial. Trials. 2021 Jan 29;22(1):104. doi: 10.1186/s13063-021-05042-w. PMID 33514408
- See also: World Health Organization. 2012. Clasificación Internacional de Enfermedades. 9a Modific. ed. Secretaría Ministerio de Sanidad, Política Social e Igualdad. Madrid. — https://www.mscbs.gob.es/estadEstudios/estadisticas/docs/CIE9MC_8ed.pdf